CLINICAL TRIAL: NCT00040625
Title: ALIMTA (Pemetrexed) Alone or in Combination With Cisplatin for Patients With Malignant Mesothelioma.
Status: Approved for marketing | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Other Study IDs: 6093; H3E-US-JMFE
Record Dates: First submitted 2002-07-02; First posted 2002-07-04 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2007-03

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Pemetrexed; Cisplatin

INTERVENTIONS:
Drug: Pemetrexed
Drug: Cisplatin

SUMMARY:
This study is to evaluate the effects (good and bad) of ALIMTA and Cisplatin or ALIMTA alone on you and your malignant pleural mesothelioma as well as make ALIMTA available to patients who qualify for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have a proven diagnosis of malignant mesothelioma in patients not candidates for curative surgery
* Prior chemotherapy for your disease is allowed
* Measurable lesion is not required
* Have a adequate performance status
* Sign an informed consent form

Exclusion Criteria:

* You are excluded from this trial if you have received any investigational agent within 4 week before enrolling in this study
* You are excluded from this trial if you have received radiation within the previous 2 weeks
* You are excluded from this trial if you are a candidates for curative surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (6):
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Basking Ridge, New Jersey, United States
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician, Porto Alegre, Rio Grande do Sul
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician, São Paulo
- Egypt (2):
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician.", Cairo
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician, Cairo
- For additional information regarding investigative sites for this trial, contact the Clinical Trials support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician, Jeddah, Saudi Arabia